CLINICAL TRIAL: NCT04029974
Title: Does the Speed of Robotic Leg Movements During Tilt-table Verticalization Affect Orthostatic Hypotension in Persons With Subacute SCI
Brief Title: Speed of Robotic Leg Movements and Orthostatic Hypotension in Subacute SCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Rehabilitation Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRC_ErigoPro_in_SCI
Record Dates: First submitted 2019-07-12; First posted 2019-07-23 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries; Orthostatic Hypotension
Keywords: Spinal cord injury; Orthostatic hypotension; Verticalization; ErigoPro; Finapres Nova
MeSH Terms: conditions — Spinal Cord Injuries; Hypotension, Orthostatic

STUDY DESIGN:
Intervention Model Description: Within-subject repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Progressive elevation (0 degrees, 25 degrees, 50 degrees, 75 degrees; x2 minutes in each position) while on robotic tilt-stepper at the cadence of 0, 40, and 80 steps/minute.
  Interventions: Device: ErigoPro

INTERVENTIONS:
Device: ErigoPro — Robotic tilt-stepper lower extremity movements at the cadence of 0, 40, and 80 steps/minute.

SUMMARY:
This study seeks to evaluate whether the speed (cadence) of lower extremity robotic movement has an impact on orthostatic hypotension and upright tolerance when training with the ErigoPro robotic tilt-stepper. It is hypothesized more frequent short-lasting leg movements (faster cadence) reduces the occurrence/severity of orthostatic hypotension better than less frequent longer-lasting leg movements (slower cadence).

DETAILED DESCRIPTION:
Orthostatic hypotension (OH) refers to a drop in blood pressure as a result of sitting up or standing up (moving against gravity). OH has been defined as a decrease in systolic (≥20 mmHg) or diastolic (≥10 mmHg) blood pressure upon transition from lying down to an upright position regardless of the presence or absence of overt symptoms (dizziness, lightheadedness, blurred vision, loss of consciousness).

OH is quite common after a spinal cord injury (SCI), especially with more severe injuries above the T6 level. OH can significantly interfere with activities of daily living and it can also interfere with participation during inpatient rehabilitation. Nearly 75% of acute SCI subjects were found to have OH and ~60% reported symptoms of OH during physical therapy activities, which limited almost 50% of the treatment sessions. Developments in rehabilitation technology have culminated in a device, a robotic tilt-stepper (RTS), e.g., known as the Erigo (Hocoma). In an RTS, the robot moves the legs through a pre-selected range of motion at different speeds to limit blood pooling during verticalization. This can be augmented by patterned functional electrical stimulation (FES), e.g., the ErigoPro.

The proof-of-principle study by the developers of the Erigo showed that passive leg movements can stabilize hemodynamic responses in healthy subjects who exhibited near-syncope when placed at 75-deg. for 30 min. Two earlier studies that examined the effect of passive leg movements on hemodynamic responses in healthy subjects used only one movement speed. Two other studies in chronic SCI (which compared the hemodynamic effects of passive leg movements alone or in combination with FES during a tilt-table verticalization) also used only one movement speed. Chi et al. showed no difference in vital signs between application of passive leg movements, FES, or the combination thereof in comparison to baseline.

Based on the literature review, it appears that no previous study has systematically examined the effects of different speeds of robotic leg movements on hemodynamic responses, which is the simplest and most user-friendly way to use RTS in a busy clinical setting. Moreover, no study recruited the most relevant target population, that is, persons with a subacute SCI who often develop OH when moved from lying down to a sitting or standing position. Therefore, it is the intent of this study to determine whether the speed of leg movement during progressive movement towards an upright position has a meaningful impact on a subjects blood pressure and onset of OH.

To test this hypothesis, healthy subjects and subjects with SCI will be recruited to participate in a one time training session with the ErigoPro. The study will occur in the SCI floor of a large rehab center. The sit-up test will be performed to assess if transitioning from supine to sitting position provokes symptoms/signs of OH. All prescribed medication will be noted and allowed as to not interfere with regular care and to reflect a real clinical practice. Each subject will then be transferred to the Erigo and secured to the device. Once secured to the device, the trial will be initiated and the subject will remain in supine for a resting period of approximately 5 minutes (to allow the subjects cardiovascular system to reach steady state) followed by another 2 minutes with their hemodynamic values continuously monitored by a beat-to-beat monitoring device (the Finapres Nova) which will aid in establishment of baseline hemodynamic thresholds. The assigned cadence (either 0, 40, or 80 steps per minute) will be initiated and the subject will then be progressed through angles of elevation including 0, 25, 50, and 75 degrees, spending approximately 2 minutes in each position with hemodynamic responses continuously monitored. If the subject demonstrates any signs/symptoms of OH or their blood pressure falls below or exceeds the established thresholds for safety or any other significant issues arise, they will be immediately returned to the supine position (0 degrees), the assigned cadence discontinued, and that portion of the trial terminated. If the subject demonstrates a return to baseline hemodynamic values within 5 - 10 minutes and they agree to continuation of the trial, they will be progressed to the next assigned speed. Should they not return to baseline values, the medical team will be contacted and the attending physician consulted. Any signs noted by the investigator or symptoms reported by the patient will be recorded and should a portion of the trial be terminated, the cause will be investigated to determine if it was truly due to OH or another issue. If the subject achieves 75 degrees for 2 minutes with no significant issues, they will be returned to supine followed by the next assigned speed being tested in the same fashion as the previously tested assigned speed.

ELIGIBILITY:
Healthy subjects and subjects with SCI:

Inclusion Criteria:

1. Reported overt signs/symptoms of OH during and/or outside of therapy sessions or primary therapist reports a drop in blood pressure consistent with OH during therapy sessions (SCI)
2. Age 16 - 70 years (Healthy & SCI)
3. Traumatic SCI AIS A - C or non-traumatic SCI, all levels of injury (SCI)
4. Time since SCI ≤ 12 weeks (SCI)
5. Weight ≤ 297 lb, leg length 29" - 39" (per ErigoPro manual) (Healthy & SCI)
6. Systolic BP >80 mmHg and <140 mmHg in supine measured by nursing staff in the 24 hours prior to recruitment. (Healthy & SCI)

Exclusion Criteria:

1. Weight bearing precautions per medical record or primary therapist report (SCI)
2. Skin lesions preventing fitting on the tilt-table or in robot cuffs (Healthy & SCI)
3. History of uncontrolled diabetes (diabetic autonomic issues) (Healthy & SCI)
4. Increase in pain/spasticity during passive leg movements during a hands-on eligibility assessment (SCI)
5. Severe fixed contractures affecting the lower limbs (hip, knee, ankle joints) (SCI)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure variation | From enrollment to end of session, approximately 2 Hours
  Systolic blood pressure will be beat-to-beat monitored. At each assigned cadence, systolic blood pressure is compared to 0-degrees elevation.

SECONDARY OUTCOMES:
Heart rate variation | From enrollment to end of session, approximately 2 Hours
  Heart rate will be beat-to-beat monitored. At each assigned cadence, heart rate is compared to 0-degrees elevation.
Frequency of orthostatic hypotension symptoms | From enrollment to end of session, approximately 2 Hours
  Subject will be instructed to report subjective symptoms (dizziness, lightheadedness, blurred vision, etc) during each elevation angle for each assigned cadence and will be prompted by open ended questions. The investigator(s) will document any additional signs of symptoms (sweating, loss of consciousness, etc) that may not have been reported by the subject.
Frequency of discontinuation of a portion of the study or termination of the entire study | From enrollment to end of session, approximately 2 Hours
  Investigator(s) will record the presence or absence of events requiring discontinuation of a portion of the study or termination of the entire study at each elevation angle for each assigned cadence.

CONTACTS AND LOCATIONS:
Overall Officials: Dobrivoje Stokic, MD, DSc, Study Director — Methodist Rehabilitation Center
Locations (1):
- Methodist Rehabilitation Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Consensus statement on the definition of orthostatic hypotension, pure autonomic failure, and multiple system atrophy. The Consensus Committee of the American Autonomic Society and the American Academy of Neurology. Neurology. 1996 May;46(5):1470. doi: 10.1212/wnl.46.5.1470. No abstract available. PMID 8628505
- [Background] Ravensbergen HJ, de Groot S, Post MW, Slootman HJ, van der Woude LH, Claydon VE. Cardiovascular function after spinal cord injury: prevalence and progression of dysfunction during inpatient rehabilitation and 5 years following discharge. Neurorehabil Neural Repair. 2014 Mar-Apr;28(3):219-29. doi: 10.1177/1545968313504542. Epub 2013 Nov 15. PMID 24243916
- [Background] Sahota IS, Ravensbergen HR, McGrath MS, Claydon VE. Cerebrovascular responses to orthostatic stress after spinal cord injury. J Neurotrauma. 2012 Oct 10;29(15):2446-56. doi: 10.1089/neu.2012.2379. Epub 2012 Sep 20. PMID 22720841
- [Background] Illman A, Stiller K, Williams M. The prevalence of orthostatic hypotension during physiotherapy treatment in patients with an acute spinal cord injury. Spinal Cord. 2000 Dec;38(12):741-7. doi: 10.1038/sj.sc.3101089. PMID 11175374
- [Background] Gillis DJ, Wouda M, Hjeltnes N. Non-pharmacological management of orthostatic hypotension after spinal cord injury: a critical review of the literature. Spinal Cord. 2008 Oct;46(10):652-9. doi: 10.1038/sc.2008.48. Epub 2008 Jun 10. PMID 18542098
- [Background] Sampson EE, Burnham RS, Andrews BJ. Functional electrical stimulation effect on orthostatic hypotension after spinal cord injury. Arch Phys Med Rehabil. 2000 Feb;81(2):139-43. doi: 10.1016/s0003-9993(00)90131-x. PMID 10668765
- [Background] Elokda AS, Nielsen DH, Shields RK. Effect of functional neuromuscular stimulation on postural related orthostatic stress in individuals with acute spinal cord injury. J Rehabil Res Dev. 2000 Sep-Oct;37(5):535-42. PMID 11322152
- [Background] Faghri PD, Yount JP, Pesce WJ, Seetharama S, Votto JJ. Circulatory hypokinesis and functional electric stimulation during standing in persons with spinal cord injury. Arch Phys Med Rehabil. 2001 Nov;82(11):1587-95. doi: 10.1053/apmr.2001.25984. PMID 11689980
- [Background] Faghri PD, Yount J. Electrically induced and voluntary activation of physiologic muscle pump: a comparison between spinal cord-injured and able-bodied individuals. Clin Rehabil. 2002 Dec;16(8):878-85. doi: 10.1191/0269215502cr570oa. PMID 12501950
- [Background] Chao CY, Cheing GL. The effects of lower-extremity functional electric stimulation on the orthostatic responses of people with tetraplegia. Arch Phys Med Rehabil. 2005 Jul;86(7):1427-33. doi: 10.1016/j.apmr.2004.12.033. PMID 16003676
- [Background] Hamzaid NA, Tean LT, Davis GM, Suhaimi A, Hasnan N. Electrical stimulation-evoked contractions blunt orthostatic hypotension in sub-acute spinal cord-injured individuals: two clinical case studies. Spinal Cord. 2015 May;53(5):375-9. doi: 10.1038/sc.2014.187. Epub 2014 Nov 4. PMID 25366533
- [Background] Chi L, Masani K, Miyatani M, Adam Thrasher T, Wayne Johnston K, Mardimae A, Kessler C, Fisher JA, Popovic MR. Cardiovascular response to functional electrical stimulation and dynamic tilt table therapy to improve orthostatic tolerance. J Electromyogr Kinesiol. 2008 Dec;18(6):900-7. doi: 10.1016/j.jelekin.2008.08.007. Epub 2008 Oct 2. PMID 18835189
- [Background] Czell D, Schreier R, Rupp R, Eberhard S, Colombo G, Dietz V. Influence of passive leg movements on blood circulation on the tilt table in healthy adults. J Neuroeng Rehabil. 2004 Oct 25;1(1):4. doi: 10.1186/1743-0003-1-4. PMID 15679913
- [Background] Yoshida T, Masani K, Sayenko DG, Miyatani M, Fisher JA, Popovic MR. Cardiovascular response of individuals with spinal cord injury to dynamic functional electrical stimulation under orthostatic stress. IEEE Trans Neural Syst Rehabil Eng. 2013 Jan;21(1):37-46. doi: 10.1109/TNSRE.2012.2211894. Epub 2012 Aug 9. PMID 22899587
- [Background] Sarabadani Tafreshi A, Riener R, Klamroth-Marganska V. Distinctive Steady-State Heart Rate and Blood Pressure Responses to Passive Robotic Leg Exercise and Functional Electrical Stimulation during Head-Up Tilt. Front Physiol. 2016 Dec 9;7:612. doi: 10.3389/fphys.2016.00612. eCollection 2016. PMID 28018240
- [Background] Claydon VE, Krassioukov AV. Orthostatic hypotension and autonomic pathways after spinal cord injury. J Neurotrauma. 2006 Dec;23(12):1713-25. doi: 10.1089/neu.2006.23.1713. PMID 17184183
- [Background] Currie KD, Wong SC, Warburton DE, Krassioukov AV. Reliability of the sit-up test in individuals with spinal cord injury. J Spinal Cord Med. 2015 Jul;38(4):563-6. doi: 10.1179/2045772315Y.0000000004. Epub 2015 Mar 4. PMID 25738545